CLINICAL TRIAL: NCT03654664
Title: A Randomized, Double-blind, Multi-center, Active-controlled, Parallel-designed, Phase III Clinical Trial to Evaluate the Immunogenicity and Safety of Inactivated Hepatitis A Vaccine in Korean Healthy Children Aged 12~23 Months
Brief Title: To Evaluate the Immunogenicity and Safety of Inactivated Hepatitis A Vaccine
Acronym: VITHA-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BR-HAV-CT-301
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Hepatitis A Vaccine
Keywords: Hepatitis A vaccine
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inactivated hepatitis A vaccine (Experimental): A 0.5ml dose is administered twice in total at an interval of 6 months to healthy children aged 12-23 months.
  Interventions: Biological: Inactivated hepatitis A vaccine
- Havrix Inj (Active Comparator): A 0.5ml dose is administered twice in total at an interval of 6 months to healthy children aged 12-23 months.
  Interventions: Biological: Havrix Inj

INTERVENTIONS:
Biological: Inactivated hepatitis A vaccine — Inactivated hepatitis A virus antigen 250 U (Name of viral strain: TZ84)
  Arms: inactivated hepatitis A vaccine
Biological: Havrix Inj — 720 ELISA/0.5 mL Junior (Inactivated hepatitis A virus antigen 160 U (Name of viral strain: HM175 Inj)
  Arms: Havrix Inj

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety after one primary dose and one additional dose of inactivated hepatitis A vaccine are administered in Korean healthy children aged 12-23 months.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the immunogenicity and safety after one primary dose and one additional dose (administered twice in total at an interval of 6 months) of inactivated hepatitis A vaccine are administered in Korean healthy children aged 12-23 months.

For this, a two-group comparison study will be conducted using a previously approved inactivated hepatitis A vaccine (Havrix Inj., manufactured by GSK) as the control vaccine to prove that the immunogenicity of the test vaccine treatment group is not inferior to the control vaccine treatment group and to statistically confirm that there is no difference in safety.

ELIGIBILITY:
Inclusion Criteria:

* A child whose parents or representative provided written consent
* A Korean child aged 12-23 months on the day of the first vaccination
* No history of hepatitis A or a having hepatitis A vaccination
* A child who was determined by the investigator that there is no problem with the participation in the clinical study according to the medical history and physical examination results

Exclusion Criteria:

* Tympanic temperature of 38℃ or above within 48 hours prior to the vaccination or on the day of vaccination
* Moderate to severe acute or chronic infectious disease on the day of vaccination
* History of sensitivity to the following drugs: neomycin, formaldehyde, gentamicin sulfate, any preventive vaccines
* Disorders in the immune system, or congenital or acquired immunodeficient diseases
* Received immunosuppressive dose of systemic corticosteroids therapy within 12weeks days before vaccination
* A child with uncontrolled epilepsy or neurological disorders
* Planned with other vaccine within 4 weeks after the vaccination date
* Administered with other vaccine within 4 weeks prior to the vaccination date
* Used immunoglobulin formulation or human plasma, or received a transfusion within 12 weeks prior to the vaccination date
* A child who has participated or is participating in another clinical trial within 12 weeks prior to the vaccination date(systemic corticosteroids administered at doses corresponding to ≤0.5 mg/kg/day of prednisolone for 14 consecutive days or less is exceptionally allowed)
* Other reasons not specified above that, in the opinion of the investigator, may make the subject ineligible to participate in the study

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | 1 month after the second administration of the investigational product
  Seroconversion criteria: Anti-HAV 20 IU/L or above

SECONDARY OUTCOMES:
Antibody titer (GMT) | 1 month after the second vaccination
  The basic statistics of the antibody titer (GMT) at 1 month after the second vaccination

OTHER OUTCOMES:
Safety endpoints Adverse events observed within 30 minutes after vaccination, solicited adverse events/adverse drug reactions, and unsolicited adverse events/adverse drug reactions through a diary, serious adverse events/adverse drug reactions, physica | Approximately 12 months after a consent to the participation
  Adverse events observed within 30 minutes after vaccination, solicited adverse events/adverse drug reactions, and unsolicited adverse events/adverse drug reactions through a diary, serious adverse events/adverse drug reactions, physical examination

CONTACTS AND LOCATIONS:
Overall Officials: HJ Cho, Study Director — BORYUNGPHARM. CO., LTD.
Locations (10):
- South Korea (10):
  - The Catholic University of Korea, Incheon St.Mary's Hospital, Incheon, Bupyeong-gu
  - The Catholic University of Korea, St.Vincent's Hospital., Suwon, Gyeonggi-do
  - Korea University Ansan Hospital, Ansan
  - Chanwon Fatima Hospital, Changwon
  - KeiMyung University Dongsan Medical Center, Daegu
  - Gachon University Gil Hospital, Incheon
  - Hanil General Hospital, Seoul
  - Korea cancer center Hospital, Seoul
  - Nowon Eulji Medical center , Eulji University, Seoul
  - Wonju Sevrance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No